CLINICAL TRIAL: NCT03378557
Title: Multicenter Prospective Registry for Periprosthetic Fractures After Hip or Knee Arthroplasty
Brief Title: Periprosthetic Fracture Registry (PPFx)
Acronym: PPFx
Status: Recruiting | Type: Observational
Sponsor: AO Innovation Translation Center (Other)
Responsible Party: Sponsor
Other Study IDs: PPFx
Record Dates: First submitted 2017-11-14; First posted 2017-12-20 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Periprosthetic Fractures; Periprosthetic Fracture Around Prosthetic Joint Implant
MeSH Terms: conditions — Periprosthetic Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This registry supports international data collection and research on PPFx treatments after hip and knee arthroplasty.

A registry such as this ultimately aims to provide far-reaching benefits to society including reduced morbidity and mortality, improved patient safety, improved quality of care and medical decision-making, reduced medical spending, and advances in orthopaedic science.

DETAILED DESCRIPTION:
To close the gap of missing clinical evidence regarding the treatment of periprosthetic fractures after arthroplasty of the hip or the knee with osteosynthesis.

To drive further study hypotheses and to answer unforeseen questions.

Main questions to be answered by the registry include (but are not exclusive) the following:

1. Influence of implants on outcome
2. Influence of surgical techniques on outcome
3. Influence of bone grafting on outcome
4. Identification of risk factors for failure
5. Identification of postoperative rehabilitation programs and its possible influence on the outcome
6. Influence of fracture type on outcome
7. To serve as a comparative dataset for future studies with improved implants and techniques

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years

  * Post-operative PPFx after total or hemi hip or total or unicondylar knee arthroplasty (including the acetabulum, femur, patella and proximal tibia) requiring

    * osteosynthesis alone or
    * component revision plus plate/nail osteosynthesis
  * Informed consent obtained, i.e.:

    * Ability of the patient or assigned representative to understand the content of the patient information / Informed Consent Form
    * Signed and dated EC / IRB approved written informed consent
  * Ability to attend post-operative follow up visits

Exclusion Criteria:

* Pregnancy or women planning to conceive within the study period
* Prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with total or hemi hip or knee arthroplasty and who have a fracture around one of the arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2018-12-31 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Classification of the fracture | Pre-operatively (Day -1)
  Classification of the fracture using the UCS and some parts of the AO/OTA fracture classification system.

SECONDARY OUTCOMES:
Fracture mechanism | Pre-operatively (Day -1)
  High / low energy trauma, pathological fracture, stem stability
Rehabilitation program | Up to 12 months
  weight bearing, bedrest, splint
Function of hip or knee | Up to 12 months
  Harris Hip Score or Knee Society score
Health related quality of life | Up to 12 months
  PROMIS pain interference and physical activity
Fracture healing | Up to 12 months
  by RUSH or RUST score
pain visual analog scale (VAS) and pain medication | Up to 12 months
  Using the pain visual analog scale (VAS) and pain medication

CONTACTS AND LOCATIONS:
Overall Officials: Karl Stoffel, MD, Principal Investigator — Universitätsspital Basel
Locations (13):
- United States (4):
  - University of Missouri Health Care, Columbia, Missouri
  - Jersey City Medical Center RWJ Barnabas Health, Jersey City, New Jersey
  - Saint Barnabas Medical Center Livingston, Livingston, New Jersey
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Universitaire Ziekenhuiven Leuven, Leuven, Belgium
- Hospital Santa Clara, Bogotá, Colombia
- Germany (3):
  - Charité Universitätsmedizin Berlin, Berlin
  - BG-Unfallklinik Ludwigshafen, Ludwigshafen
  - Universitätsklinikum Münster, Münster
- Hospital Universitario Son Llàtzer, Palma de Mallorca, Spain
- Switzerland (3):
  - Universitätsspital Basel, Basel
  - Kantonspital Baselland, Liestal
  - Universitätsspital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Uzoigwe CE, Watts AT, Briggs P, Symes T. Periprosthetic Femoral Fractures-Beyond B2. J Am Acad Orthop Surg Glob Res Rev. 2024 Aug 6;8(8):e23.00135. doi: 10.5435/JAAOSGlobal-D-23-00135. eCollection 2024 Aug 1. PMID 39110721